CLINICAL TRIAL: NCT00857064
Title: Subjective Well Being of Schizophrenic Patients in Greece
Acronym: AURA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Pontikis Panagiotis, MD Medical and Regulatory Affairs Director, AstraZeneca, SA Greece
Other Study IDs: NIS-NGR-DUM-2008/2
Record Dates: First submitted 2009-03-03; First posted 2009-03-06 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; antipsychotics; social functioning; subjective well being; Patients suffering from Schizophrenia
MeSH Terms: conditions — Schizophrenia; Social Adjustment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-interventional study aiming to provide data on the subjective effects of antipsychotic medication assessing subjective well-being and global functioning of patients with Schizophrenia under antipsychotic medication. Moreover it aims to assess their adherence to the treatment and will investigate whether there is any correlation of these factors with the clinical condition of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Diagnosis of schizophrenia according to DSM-IV
* The patient must have been prescribed an atypical antipsychotic for at least 4 weeks before the first study visit

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target Group:Patients suffering from Schizophrenia treated in private practice
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Subjective well being | Relative score reported in SWBN scale at the visit. No baseline comparison
Assessment of functioning | Relative score reported in GAF scale at the visit. No baseline comparison

SECONDARY OUTCOMES:
Assessment of Compliance to therapy | Relative score reported in BARS scale at the visit. No baseline comparison
Assessment of General Psychopathology | Relative score reported in PANNS scale at the visit. No baseline comparison
Assessment of Clinical Condition | Relative score reported in CGIS scale at the visit. No baseline comparison

CONTACTS AND LOCATIONS:
Overall Officials: Errikos Tzempelikos, Dr, Principal Investigator — Sismanoglio Hospital, Psychiatric Department, Greece
Locations (24):
- Greece (24):
  - Research Site, Agrinio
  - Research Site, Alexsandroupoli
  - Research Site, Argos
  - Research Site, Arta
  - Research Site, Athens
  - Research Site, Crete
  - Research Site, Drama
  - Research Site, Edessa
  - Research Site, Elefsina
  - Research Site, Giannitsá
  - Research Site, Ioannina
  - Research Site, Karditsa
  - Research Site, Katerini
  - Research Site, Kavala
  - Research Site, Kozani
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Piraeus
  - Research Site, Preveza
  - Research Site, Rhodes
  - Research Site, Serres
  - Research Site, Thebes
  - Research Site, Thessaloniki
  - Research Site, Volos